CLINICAL TRIAL: NCT00201929
Title: Development and Evaluation of Different Versions of the Decision Board for Early Breast Cancer
Brief Title: A Decision Aid for Women With Early Stage Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); Supportive Cancer Care Research Unit (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SCCR-Unit-Decision Board; DAMD17-98-1-8100
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2007-06-29 (Estimated); Status verified 2007-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; decision aid; Decision Board; information transfer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Procedure: Standard Decision Board
Procedure: Computer Decision Board
Procedure: Paper Decision Board

SUMMARY:
To enhance information transfer and decision making for women with breast cancer.

DETAILED DESCRIPTION:
Our specific objectives are: (i) to develop computer and paper based versions of the Decision Boards for (a) chemotherapy for early stage breast cancer (chemotherapy versus no treatment), (b) mastectomy versus lumpectomy plus radiation and (ii) to compare the relative effectiveness of the computer and paper based versions with the standard Decision Board for patients with early breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Chemotherapy Group:

* Female
* Histologically documented invasive carcinoma of the breast treated with modified radical mastectomy or lumpectomy
* Axillary node dissection
* Chemotherapy alone or in addition to tamoxifen as an appropriate treatment option

Surgery Group:

* Female
* Newly diagnosed carcinoma of the breast diagnosed either by cytology or pathological examination, OR if no biopsy, a strong clinical suspicion of malignancy
* Clinical stage I or II disease
* Candidate for breast conserving surgery

Exclusion Criteria:

Chemotherapy Group:

* Candidate for CEF chemotherapy
* Clinical evidence of metastatic disease
* Serious comorbidity that would preclude receiving chemotherapy treatment
* Unable to speak or read English fluently (including visual impairment)
* Mentally incompetent including any psychiatric or addictive disorders that would preclude shared decision-making

Surgery Group:

* Previous surgery for breast cancer
* Previous breast irradiation
* Pregnant
* Clinical suspicion of bilateral breast cancer
* Serious comorbidity that would preclude definitive surgery
* Unable to speak or read English fluently (including visual impairment)
* Mentally incompetent including any psychiatric or addictive disorder that would preclude shared decision making

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2002-04; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Patient comprehension
Patient satisfaction with information transfer

SECONDARY OUTCOMES:
Patient satisfaction with decision making
Physician satisfaction with information transfer
Physician satisfaction with decision making
Time required for administration of the instrument
Patient preference for decision making

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Whelan, MD, Study Chair — Juravinski Cancer Centre
Locations (9):
- Canada (9):
  - Denise Schnider, Brantford, Ontario
  - Ken Reed, Guelph, Ontario
  - Susan Reid, Hamilton, Ontario
  - Barbara Heller, Hamilton, Ontario
  - Ken Sanders, Hamilton, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Nabih Mattar, Simcoe, Ontario
  - Anna Kobylecky, St. Catharines, Ontario
  - Peter Koziarz, Welland, Ontario